CLINICAL TRIAL: NCT06846333
Title: Effect of Opioid-free Anesthesia Protocol on Quality of Recovery After Major Surgery in Geriatric Patients
Brief Title: Opioid-free Anesthesia and Quality of Recovery After General Anesthesia
Status: Not yet recruiting | Type: Observational
Sponsor: Selcuk University (Other)
Responsible Party: Principal Investigator, Meltem Mavuş, MD, Selcuk University
Other Study IDs: 2025/2
Record Dates: First submitted 2025-02-03; First posted 2025-02-26 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-02

CONDITIONS: Opioid-free Anesthesia; Geriatric Population

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Opioid-Based Anesthesia (Group 1): Group I patients underwent induction with propofol (2.0 mg/kg), fentanyl (2 µg/kg), and rocuronium (0.6 mg/kg). Maintenance of anesthesia was achieved using remifentanil (0.1-0.25 µg/kg/min), titrated to maintain a BIS level of 40-60, and the inhalation anesthetic agent sevoflurane, targeting a MAC of 1.0-1.5. No external intervention was made regarding drug dosages
- Opioid-Free Anesthesia (Group 2): Group II patients underwent induction with propofol (2.0 mg/kg), ketamine (0.3 mg/kg), and rocuronium (0.6 mg/kg). Maintenance of anesthesia was achieved using ketamine (10-45 µg/kg/min), titrated to maintain a BIS level of 40-60, and sevoflurane, targeting a MAC of 1.0-1.5. In Group II, the ketamine infusion was discontinued 30 minutes before the end of the surgery. No external intervention was made regarding drug dosages.

SUMMARY:
This study aimed to evaluate the effect of an opioid-free anesthesia protocol on postoperative recovery quality in patients aged 65 years and older undergoing major surgery. Recovery quality was assessed using the Quality of Recovery-15 (QoR-15) questionnaire. Findings are expected to contribute to optimizing anesthesia practices in the elderly population by improving recovery quality and reducing opioid-related side effects.

DETAILED DESCRIPTION:
This prospective observational study aims to evaluate the impact of an opioid-free anesthesia (OFA) protocol on postoperative recovery quality in geriatric patients aged 65 years and older undergoing major non-cardiac surgery. Recovery quality will be assessed using the Quality of Recovery-15 (QoR-15) questionnaire at 24, 48, and 72 hours postoperatively. Secondary outcomes include postoperative pain intensity (measured via VAS), opioid consumption (measured through patient-controlled analgesia devices), the incidence of postoperative cognitive dysfunction (POCD) assessed using the Mini-Mental Test (MMT) and the Clock Drawing Test, and the frequency of opioid-related adverse events (nausea, vomiting, constipation, urinary retention, dizziness, and others). Furthermore, intraoperative hemodynamic stability, extubation time, time to spontaneous ventilation recovery, and lengths of stay in the post-anesthesia care unit (PACU) and the hospital will also be recorded.

The rationale for this study is rooted in the significant side effects of opioids, such as postoperative nausea and vomiting (PONV), hyperalgesia, sedation, and respiratory depression, which can prolong recovery time and hospital discharge. To accelerate postoperative recovery and minimize opioid-related side effects, "Enhanced Recovery After Surgery (ERAS)" protocols, which have gained popularity in recent years, include OFA as an alternative analgesic strategy. OFA protocols provide multimodal analgesia through non-opioid drugs and techniques targeting various pain pathways, potentially reducing the incidence of chronic pain and expediting recovery.

A key component of the OFA protocol used in this study is ketamine, which has shown efficacy in reducing neuroinflammation and improving cognitive function, making it particularly relevant in the elderly population at risk of postoperative cognitive dysfunction. While evidence supporting the benefits of OFA in various surgical fields such as gynecology, orthopedics, and gastrointestinal surgeries is growing, there remains a lack of data on its effects on recovery outcomes in geriatric patients undergoing major surgeries. This study aims to address this gap by providing comprehensive data on the impact of OFA on recovery quality, opioid-related adverse events, and perioperative outcomes in this vulnerable population.

Patients will be divided into two groups based on the anesthesiologist's clinical preference:

1. Opioid-Based Anesthesia (Group 1): Induction with propofol, fentanyl, and rocuronium; maintenance with remifentanil and sevoflurane.
2. Opioid-Free Anesthesia (Group 2): Induction with propofol, ketamine, and rocuronium; maintenance with ketamine and propofol infusions, along with sevoflurane.

Both groups will undergo standard perioperative monitoring, including BIS (bispectral index) for anesthesia depth and continuous hemodynamic monitoring. Recovery parameters such as extubation time, spontaneous ventilation recovery, and PACU length of stay will be recorded in detail. Postoperatively, the QoR-15 questionnaire will be completed at 24, 48, and 72 hours, with follow-up by telephone for patients discharged early.

This study is expected to contribute to the limited literature on the application of OFA in geriatric surgical patients. By highlighting the potential benefits of OFA in enhancing postoperative recovery, reducing opioid consumption, and preventing opioid-related adverse events, this research aims to provide insights for safer and more effective anesthesia practices in the elderly population.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 65 and older
* Undergoing major elective non-cardiac surgery under general anesthesia
* Classified as ASA I-II-III
* With sufficient cognitive ability to complete a questionnaire were included in the study

Exclusion Criteria:

* Patients requiring rapid sequence induction for emergency cases
* Those with severe psychiatric or cognitive disorders preventing questionnaire evaluation
* A body mass index < 18 or > 39 kg/m²
* Allergy or contraindication to any drug included in the study
* A history of chronic pain or chronic opioid use
* Uncontrolled epilepsy, decompensated heart failure
* Chronic kidney or liver failure
* Preoperative bradycardia with atrioventricular block (2nd or 3rd degree)
* Heart rate < 50 bpm due to chronic beta-blocker therapy
* Those using medications that prolong the QT interval
* Patients whose anesthesia regimen was intraoperatively changed (from opioid-free to opioid-containing anesthesia)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Geriatric patients over 65 years old undergoing major surgery
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-02-20 (Estimated); Primary Completion 2025-04-25 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Quality of Recovery | The quality of recovery will be assessed using the QoR-15 scale at 24, 48, and 72 hours postoperatively.
  The quality of recovery will be evaluated using the quality of recovery 15 (QoR-15) scale.QoR-15 is a 15-item questionnaire that assesses the patient's emotional state, physical comfort, psychological support, physical independence, and pain status, with each question scored between 0 (never) and 10 (always); a total score of less than 90 is considered poor, a score between 90 and 121 is moderate, a score between 122 and 135 is good, and a score above 135 indicates excellent recovery.

SECONDARY OUTCOMES:
Postoperative cognitive dysfunction | Postoperative cognitive dysfunction will be evaluated using the MMSE, administered preoperatively and at 24 hours postoperatively.
  Postoperative cognitive dysfunction will be evaluated using the Mini Mental State Examination (MMSE). The MMSE score is considered to indicate normal cognitive function if it ranges between 30 and 24, mild cognitive impairment if it is between 23 and 20, moderate cognitive impairment if it falls between 19 and 10, and severe cognitive impairment if it is 9 or below.
Postoperative cognitive dysfunction | Postoperative cognitive dysfunction will be evaluated using the Clock Drawing Test, administered preoperatively and at 24 hours postoperatively.
  Postoperative cognitive dysfunction will be evaluated using the Clock Drawing Test. According to the Clock Drawing Test, a score between 8 and 10 indicates normal cognitive function, a score between 5 and 7 suggests mild cognitive impairment, and a score of 4 or below signifies moderate to severe cognitive impairment.
Postoperative pain management | Postoperative pain will be assessed using the Visual Analog Scale (VAS) at PACU, and at 6, 12, 24, and 48 hours postoperatively.
  Postoperative pain assessment will be evaluated using the Visual Analog Scale (VAS). VAS is a subjective and visual assessment method where the patient rates pain intensity on a scale from 0 (no pain) to 10 (worst pain).
Opioid consumption | The total drug consumption and the amounts administered via the PCA device at postoperative 6, 12, 24, and 48 hours will be recorded.
  Opioid consumption will be evaluated using Contramal via a patient-controlled analgesia (PCA) device.
To evaluate recovery profile | The time to spontaneous ventilation, defined as the time between the cessation of anesthesia and the initiation of spontaneous ventilation, was recorded in seconds during the perioperative period.
  The time elapsed until spontaneous ventilation (the period between the cessation of anesthesia and the initiation of spontaneous ventilation) was recorded in seconds.
To evaluate recovery profile | The extubation time, defined as the time from the cessation of anesthesia to extubation, was recorded in seconds during the perioperative period.
  Time to extubation time (the time between anesthetic discontinuation and extubation) was recorded in seconds.
To evaluate recovery profile | The eye-opening time, defined as the time between the cessation of anesthesia and eye opening in response to verbal or painful stimuli, was recorded in seconds during the perioperative period.
  The eye-opening time during the perioperative period (the time between anesthetic discontinuation and eye opening in response to verbal stimulus or painful pinching) was recorded in seconds.
To evaluate recovery profile | The time to discharge from the PACU was recorded in minutes, defined as the time from arrival at the PACU to transfer to the ward during the perioperative period.
  The PACU discharge time (the time from arrival at the PACU to transfer to the ward) was recorded in minutes.
To evaluate recovery profile | The length of hospital stay was recorded in days during the perioperative period, calculated by subtracting the admission date from the discharge date
  The length of hospital stay (calculated by subtracting the admission date from the discharge date) was recorded in days.
Opioid-Related Adverse Events | Opioid-related adverse events observed within 72 hours after surgery were recorded.
  Opioid-related adverse events (nausea, vomiting, constipation, difficulty urinating, difficulty concentrating, drowsiness or difficulty staying awake, dizziness, feeling sleepy, general fatigue or weakness, itching, dry mouth, and headache).